CLINICAL TRIAL: NCT05401578
Title: Canakinumab for the Treatment of Postprandial Hypoglycemia - CanpHy Study
Brief Title: Canakinumab for the Treatment of Postprandial Hypoglycemia
Acronym: CanpHy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02325; kt21Donath2
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Postprandial Hypoglycemia
Keywords: bariatric surgery; IL-1 receptor antagonist; postbariatric hypoglycemia; canakinumab; quality of life
MeSH Terms: conditions — Hypoglycemia | interventions — canakinumab

STUDY DESIGN:
Intervention Model Description: National, multicenter, 1:1 randomized, placebo-controlled, parallel-group, double-blind superiority trial
Who Masked: Participant, Investigator
Masking Description: Both subjects and investigators will be blinded. A nurse independent of the research group will be responsible for treatment blinding and preparation of trial drugs throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Intervention: Canakinumab (Active Comparator): Standard dose of canakinumab (Ilaris®; Novartis Switzerland), i. e. 150 mg subcutaneously.
  Canakinumab (Ilaris®, Novartis) is a recombinant, human monoclonal IgG1/kappa antibody inhibiting IL-1β by neutralizing its biological activity through binding to the IL-1 receptor.
  Interventions: Drug: Canakinumab
- Control Intervention: Placebo (0.9% NaCl) (Placebo Comparator): Placebo: 1 ml of 0.9 % NaCl
  Interventions: Drug: Placebo (0.9% NaCl)

INTERVENTIONS:
Drug: Canakinumab — Canakinumab (Ilaris®, Novartis Switzerland) will be used in the recommended standard dose of 150 mg subcutaneously once. Patients will be randomized at visit 2 = Baseline to either placebo (1 ml 0.9 % saline solution s.c.) or treatment with 1 ml 150 mg canakinumab solution s.c. in a 1:1 manner.
  Arms: Study Intervention: Canakinumab
Drug: Placebo (0.9% NaCl) — 1 ml 0.9 % saline solution s.c. Patients will be randomized at visit 2 = Baseline to either placebo (1 ml 0.9 % saline solution s.c.) or treatment with 1 ml 150 mg canakinumab solution s.c. in a 1:1 manner.
  Arms: Control Intervention: Placebo (0.9% NaCl)

SUMMARY:
The primary objective of this randomized trial is to test whether a treatment with canakinumab is superior to placebo in patients with postprandial hypoglycemia after bariatric surgery, that is if it improves health related quality of life (mentally or physically) or reduces the risk of hypoglycemic events.

DETAILED DESCRIPTION:
Postprandial hypoglycemia is a debilitating medical complication after bariatric surgery for which no approved pharmacological treatment exists. In a former study, the IL-1 receptor antagonist Anakinra statistically significantly reduced the number of symptomatic hypoglycemia.

This randomized clinical trial is to directly evaluate clinical outcomes and patient-relevant benefits of treatment with the IL-1 receptor canakinumab over 28 days. The primary objective of this randomized trial is to test whether a treatment with canakinumab is superior to placebo in patients with postprandial hypoglycemia after bariatric surgery, that is if it improves health related quality of life (mentally or physically) or reduces the risk of hypoglycemic events.

For each subject, a maximum study duration of four months is anticipated with: screening visit 1 (1 h), screening phase (10-day screening phase for postprandial hypoglycemia using a blinded continuous glucose monitoring system (CGMS, Dexcom G6)), randomization/starting visit (visit 2, 1.5 h) followed by a 28 days intervention period with two additional study days (visit 3 and 4, 0.5 h, change of blinded continuous glucose monitoring system (CGFS sensor), diary documentation, adverse events) and end of treatment visit (visit 5). A follow-up visit will be done two months after the end of the treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients after bariatric surgery (i.e. sleeve gastrectomy, Roux-en-Y gastric bypass, omega-loop bypass, biliopancreatic diversion) with documented hypoglycemia, i. e. < 3.0 mmol/l and at least 5 hypoglycemic episodes per week despite dietary modification
* For women with child-bearing potential, willingness to use contraceptive measures adequate to prevent pregnancy during the study
* Informed Consent as documented by signature

Exclusion Criteria:

* Any type of diabetes mellitus according to ADA criteria
* Intolerance to the study drug
* Signs of current infection
* Any use of immunosuppressive medication
* Use of any drug therapy for postbariatric hypoglycemia apart from acarbose (all remaining drugs have to be discontinued four half-life times before screening phase)
* Neutropenia (leukocyte count < 1.5 × 109/L or ANC < 0.5 × 109/L)
* Anemia (hemoglobin < 11 g/dL for males, < 10 g/dL for females)
* Clinically significant kidney or liver disease (creatinine > 1.5 mg/dL, AST/ALT > 2 × ULN, alkaline phosphatase > 2 × ULN, or total bilirubin [tBili] > 1.5 × ULN)
* Uncontrolled congestive heart failure
* Uncontrolled malignant disease
* Currently pregnant or breastfeeding
* Known or suspected non-compliance, drug or alcohol abuse
* Meeting the criteria for vulnerability (e.g. participants incapable of judgment or participants under tutelage)
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another clinical trial using investigational drugs in the last 30 days or planned participation in the next 60 days
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Health related quality of life (mental health) | At Baseline (study day 1), day 29 (-1 /+2 days) and at Follow- up (day 90 +/- 11 days)
  Health related quality of life (mental health; as assessed by the SF-36 mental health component score; MCS). The lower the score the more disability.
Change in Health related quality of life (physical health) | At Baseline (study day 1), day 29 (-1 /+2 days) and at Follow- up (day 90 +/- 11 days)
  Health related quality of life (physical health; as assessed by the SF-36 physical component score; PCS). The lower the score the more disability.
Number of Hypoglycemic events | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Hypoglycemic events defined as glucose values below 3.0 mmol/l

SECONDARY OUTCOMES:
Change in Postprandial Symptoms of hypoglycemia according to Edinburgh Hypoglycemia Scale (EHSS) | At Baseline (study day 1), day 29 (-1 /+2 days) and at Follow- up (day 90 +/- 11 days)
  Postprandial Symptoms of hypoglycemia defined as acute onset of typical symptoms according to Edinburgh Hypoglycemia Scale. The EHSS is an instrument to evaluate patients' experiences of symptoms in a typical hypoglycemic episode. It comprises 11 symptoms divided into three domains-neuroglycopenic, autonomic, and malaise, which are evaluated by a 7-point Likert scale "1= Not at all, 7= Very severely". The postprandial period is defined as 3 hours following meal intake.
Change in Hypoglycemia unawareness (measured by modified Clarke Score) | At Baseline (study day 1), day 29 (-1 /+2 days) and at Follow- up (day 90 +/- 11 days)
  The Clarke questionnaire consists of eight specific items characterizing awareness of hypoglycemia giving a total score of "0" to "7 (score ≥4 suggests inadequate hypoglycemia awareness; a score ≤2 suggests normal hypoglycemia awareness
Change in Fear of hypoglycemia (measured on a scale of 0 to 10) | At Baseline (study day 1), day 29 (-1 /+2 days) and at Follow- up (day 90 +/- 11 days)
  The fear of hypoglycemia will be assessed by using a 10-cm long visual analogue scale graded from "0 - no fear at all" to "10 - massive fear"
Time below range (TBR; % of sensor glucose readings and time between 3.0 and 3.8 mmol/L) | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Time below range (TBR; % of sensor glucose readings and time between 3.0 and 3.8 mmol/L)
Time in hypoglycemia: % of sensor glucose readings and time below 3.0 mmol/L | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Time in hypoglycemia: % of sensor glucose readings and time below 3.0 mmol/L
Pattern of sensor glucose | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Pattern of sensor glucose, defined as the slope of postprandial increase (calculated as the maximal rate of increase observed over 20min in the postprandial period) and decrease CanpHy-Study Version 1.2 of date 02.04.2022 Page 26 of 47 (calculated as the maximal rate of decrease over 20min in the postprandial period). The postprandial period is defined as 3 hours following meal intake.
Glycemic variability (defined as the coefficient of variation (CV) of sensor glucose) | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Glycemic variability (defined as the coefficient of variation (CV) of sensor glucose)
Mean amplitude of sensor glucose excursions (MAGE) | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Mean amplitude of sensor glucose excursions (MAGE)
Change in Body weight | From Baseline (study day 1) to day 29 (-1 /+2 days)
  Change in Body weight
Total adverse events | From Baseline (study day 1) to Follow- up (day 90 +/- 11 days)
  Total adverse events
Serious adverse events | From Baseline (study day 1) to Follow- up (day 90 +/- 11 days)
  Number of Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marc Y Donath, Prof. Dr., Principal Investigator — University of Basel
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Division of Endocrinology, Diabetes and Metabolism, Basel
  - Cantonal Hospital Olten, Division of Endocrinology, Olten

IPD SHARING:
Plan to Share IPD: No
Results will be published in a relevant scientific journal and communicated to participants and relevant institutions through dissemination activities. Individual data are accessible on request.